CLINICAL TRIAL: NCT06440057
Title: A Phase I Dose Escalation Study of Tolerability, Safety, Efficacy, and Pharmacokinetics of ZG006 in Participants With Advanced Small Cell Lung Cancer or Neuroendocrine Carcinoma, Followed by a Phase II Dose Expansion Study in Participants With Neuroendocrine Carcinoma.
Brief Title: Dose Escalation Study of ZG006 in Participants With Advanced Small Cell Lung Cancer or Neuroendocrine Carcinoma, Followed by Dose Expansion Study in Participants With Neuroendocrine Carcinoma.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG006-003
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): A total of six dose escalations were preset: 0.1 mg, 0.3 mg, 1 mg, 3 mg.
  Interventions: Biological: ZG006
- Dose Expansion (Experimental): Participants will receive the RP2D identified in Dose Escalation Study .
  Interventions: Biological: ZG006

INTERVENTIONS:
Biological: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.

SUMMARY:
This is a multicenter, open-label phase I/II study, divided into 2 parts:

Part 1 involves a dose-escalation study of ZG006 in which the safety and tolerability of ZG006 in patients with advanced small cell lung cancer or neuroendocrine carcinoma are explored. Upon completion of Part 1, investigators and the sponsor will discuss and determine two recommended phase II doses (RP2D) based on safety, preliminary efficacy, and pharmacokinetic results for use in Part 2.

Part 2 is a phase II dose-expansion study of ZG006, aiming to investigate the efficacy and safety of ZG006 in patients with Neuroendocrine Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form;
* Male or female 18~75 years of age;
* Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1;
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Participants were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants achieving a confirmed complete response (CR) or partial response(PR) based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 2 years
  The types and frequencies of adverse events (AEs) evaluated according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No